CLINICAL TRIAL: NCT06829550
Title: 3D Scanning as an Advanced Tool for Identifying Tooth Lesions in Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Aline Rogeria Freire de Castilho, Principal Investigator, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24373
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries in Children; Tooth Erosion; Fluorosis, Dental; Dental Caries
Keywords: scanning for dental problems; computer-assisted image processing; tooth wear; dental fluorosis; intraoral scanner; dental caries; dental decay; tooth erosion
MeSH Terms: conditions — Tooth Erosion; Fluorosis, Dental; Dental Caries; Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- direct- visual examination and indirect- 3D digital scanning (Other): Two diagnostic methods (direct- visual examination and indirect- 3D digital scanning) will be conducted for each participant (n=30), comparing their effectiveness in detecting dental caries, erosive tooth wear, and fluorosis.
  Interventions: Diagnostic Test: indirect- 3D digital scanning

INTERVENTIONS:
Diagnostic Test: indirect- 3D digital scanning — examination for dental caries, erosive tooth wear and dental fluorosis using direct assessment (visual) and indirect assessment (digital scanning)

SUMMARY:
This study focuses on assessing dental caries, erosive tooth wear, and fluorosis in primary teeth using a 3D intraoral digital scanner. The investigator will validate findings using three key indices: ICDAS (for caries), BEWE (for erosive wear), and TF (for fluorosis). Teeth will be cleaned and examined visually using dental tools and light. After visual checks, teeth will be scanned with a 3D intraoral scanner. Children aged 3-12 years with fully erupted primary teeth, seeking dental treatment at the Department of Pediatric Dentistry, Indiana University School of Dentistry.

The visual examination and digital scanning will be performed just once and during the dental appointment at the clinic of Pediatric Dentistry following the protocols used in the clinical routine. It is expected to complete the visual examination and the digital scanning in 30 minutes.

DETAILED DESCRIPTION:
Experimental design: This study is based on information obtained in a pilot study in the framework of a "validation study" previously to an in vivo study. Investigators will be trained in 3 different indices to register and grade the lesions to obtain reproducible data. International caries detection and assessment system (ICDAS - Pitts et al., 2013), Basic Erosive Wear Examination (BEWE - Schlueter et al., 2020), and TF index (Thylstrup & Fejerskov, 1978) will be used for detection of caries lesions, erosive tooth wear, and dental fluorosis, respectively.

Patient recruitment: The research protocol was approved by the Institutional Review Board (# 24373). After IRB approval and previous to any intervention, a signed informed consent form will be obtained from the legal guardians of each child. Children aged between 3 and 12 years old, presenting any fully erupted primary teeth, searching for dental treatment at the Department of Pediatric Dentistry, Indiana University School of Dentistry will be included in this study.

Visual examination: Before visual examination, teeth will be cleaned using a bristle brush, prophylaxis paste and mirror, washed, and carefully air dried. Isolator will be used to control the saliva during the prophy. For the index detection using the visual examination of the different indices on each tooth's, the primary upper and lower incisors, canines and molars will be dried with compressed air, and each tooth's buccal, palatal/lingual, and occlusal surfaces will be examined visually using adequate dental instruments for each index. A headlight or overhead/dental unit light will be directly over the teeth. The diagnosis of caries lesions, erosive tooth wear, and dental fluorosis will be carried out separately. ICDAS, BEWE, and TF systems will be registered and graded the lesions according to table 1. Once the visual examination is completed, the data will be stored to be compared with intraoral scanner later.

Digital scanning: After completing the visual examination, the investigators will be calibrated using 3Shape TRIOS 4 intraoral scanner and 3Shape Unite software for data processing according to the manufacturer's instructions. The primary teeth's buccal, palatal/lingual, and occlusal surfaces will be scanned with a 3D intraoral scanner (IOS) (TRIOS 4; 3Shape A/S, Copenhagen, Denmark) and register with a number. There will be no headlight or overhead/dental unit light directly over the teeth to be scanned. Subsequently, using the 3Shape Unite software, each tooth will be analyzed separately on all its surfaces (as with the visual examination, the ICDAS, BEWE, and TF, indices will be detected) by using the 3Shape software and an entire screen of a 15.5" Dell laptop. Following, the 3D image will be magnified until only lesion can be seen and each surface will be observed systematically for each index.

ELIGIBILITY:
Inclusion Criteria:

Children aged between 3 and 12 years old, presenting at least one fully erupted primary tooth.

Exclusion Criteria:

* Unerupted primary teeth.
* Restored teeth.
* Children under 3 or older than 12 years old.
* Children using medication.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate caries using intraoral digital scanning | Evaluation will occur during the single 1 day visit
  Dental caries - detection of caries lesions in primary teeth comparing the use of intraoral digital 3D scanning (imaging) to a traditional clinical exam
Evaluate Erosive tooth wear using digital scanning | Evaluation will occur during the single 1 day visit
  Erosive Tooth Wear - detection of erosive tooth wear patterns in primary teeth comparing the use of intraoral digital 3D scanning (imaging) with a traditional clinical erosion tooth wear exam
Evaluate fluorosis using intraoral digital scanning | Evaluation will occur during the single 1 day visit
  Fluorosis: - detection of fluorosis in primary teeth comparing the use of intraoral digital 3D scanning (imaging) with a traditional clinical fluorosis exam

CONTACTS AND LOCATIONS:
Overall Officials: Aline Castilho, DDS, Principal Investigator — Indiana Unviersity
Locations (1):
- Indiana University School of Dentistry (IUSD), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No